CLINICAL TRIAL: NCT04466644
Title: A Multicenter, Prevalence Study to Evaluate the Infectious and Immunological Status of COVID-19 in Asymptomatic Subjects Attending ART Centres After the Pandemic Lockdown in the USA
Brief Title: COVID-19: A Prevalence Study of Two ART Centres After the Pandemic Lockdown in the USA (COVID-19 Free Clinics)
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX2-COV-JC-20-04; 20201490 (Other: Western IRB Tracking Number)
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood
  * Saliva
  * Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The regulars of IVF clinics in the USA: Mainly asymptomatic individuals composed by patients who are attending their regular medical consultation and/ clinic staff of the participant sites, located in two areas of the USA with different pandemic status, and undergoing PCR and ELISA tests for diagnosis of COVID-19 before initiating the work after the lockdown.
  Interventions: Diagnostic Test: ELISA; Diagnostic Test: RT-PCR

INTERVENTIONS:
Diagnostic Test: ELISA — Antibody test (serology) in the blood samples to determine if the subject was previously infected.
Diagnostic Test: RT-PCR — For detecting the presence of SARS-CoV-2 RNA molecule in the nasopharyngeal swabs and saliva.

SUMMARY:
In late December 2019, a new coronavirus strain emerged causing coronavirus disease 2019 (COVID19). Since then, COVID19 has become a global pandemic outbreak being declared a "public health emergency of international concern" by the International Health Regulations Emergency Committee of the WHO on January 30, 2020. Several emergency measures have been implemented in different countries such as lockdown, social distancing, and testing.

The pandemic concerns to public worldwide but also to couples aiming to conceive through natural means or undergoing assisted reproductive technologies (ART). The American Society of Reproductive Medicine (ASRM) as well as European Society of Human Reproduction and Embryology (ESHRE) have recommend a precautionary approach and advise that all fertility patients considering or planning treatment, even if they do not meet the diagnostic criteria for COVID-19 infection, should avoid becoming pregnant at this time until more is known about the virus. Therefore, new cycles for infertility patients as well as non-medically urgent gamete preservation treatments, such as social egg freezing, have been suspended deferring embryo transfer in those patients with initiated cycles. In this moment, when reopening phases are being undertaken in most countries, the decision to resume the In vitro fertilization (IVF) treatment in a safe environment to the healthcare workers and patients is the biggest concern of the ART clinics.

The present study aims to describe the percentage of COVID-19 condition (naïve, immune, and currently infected) in asymptomatic individuals from two different ART centres. For this purpose, the ART centres' personnel and patients will be tested for COVID-19 before resume the clinic daily routine just after the lockdown period.

DETAILED DESCRIPTION:
On March 11th 2020, WHO characterized COVID-19 as a pandemic and on March 13th, the President of the United States declared the COVID-19 outbreak a "national emergency". In order to fight this pandemic, emergency measures have been implemented in different countries such as lockdown, social distancing and testing. It is known that these measures have differed among countries and due to the lack of tests worldwide, the real number of affected and/or immunized people remains largely unknown. In this context, the daily most important surrogate markers have been the numbers of infected hospitalized and deceased population. However, asymptomatic infections are not uncommon (representing up to 30% of infected cases) and the detection of this population seems crucial to prevent their potential transmission and to guide the development of measures to control the ongoing pandemic.

This is a descriptive, prevalence study that aims to define the current contagious risk and immune status to SARS-CoV-2/COVID-19 infection in two reproduction health centers in the USA located in Utah and Massachusetts. Aiming for the better technical procedures available, different biological samples (nasopharyngeal swab, saliva, and blood sample) from each participant will be tested applying two different methodologies already approved by Health Authorities, and nowadays the most commonly used for the COVID-19 diagnose: Reverse Transcriptase - Polymerase Chain Reaction (RT-PCR) for the analysis of the nasopharyngeal swabs and saliva samples and Immunoassay by serology for the blood serum analysis.

A total of 400 participants, distributed equally between the two participant centers, are expected to be included in 2 months.The total expected duration of the study is 4 months for collecting, processing and analysing samples from participants (patients and clinical staff), although the participation in the study will entail just a single visit (coinciding with the same day of the samples collection). After that visit, no further interventions or follow-up directly related to this study will be required.

Data exported from the clinical histories and source documents will be duly codified to protect the clinical and personal information of patients in accordance with the current legislation. This information will be exported to an electronic Case Report Form (eCRF) for its analysis. Given the exceptional situation that the world is facing with the COVID-19 pandemic, U.S. authorities demand the report of all tested cases, so patient´s data will be communicated to the U.S. national health authorities when the result of the test is positive.

ELIGIBILITY:
Inclusion Criteria:

* Age of majority subjects whose written informed consent approved by the IRB has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* Site staff who are re-incorporating to the centers and patients who are attending their medical appointment for their regular IVF treatment.
* Mainly asymptomatic individuals from the ART clinics, before initiating the work right after the lockdown period.

Note: COVID-19 symptomatology may appear 2-14 days after exposure to the virus and may include at least one of the following symptoms:

* Fever
* Cough
* Shortness of breath or difficulty breathing
* Chills
* Repeated shaking with chills
* Muscle pain
* Headache
* Sore throat
* New loss of taste or smell

Exclusion Criteria:

• Not applicable as there is not exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mainly asymptomatic subjects composed by patients who are attending for their regular medical consultation and clinic staff for COVID-19 infection from the two participant sites, located in two areas with different pandemic status, before initiating the work immediately after the lockdown period.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of contagiousness in asymptomatic individuals by PCR with nasopharyngeal swabs | 2 months
  Statistical quantification of the prevalence of contagiousness in asymptomatic individuals attending IVF clinics in the USA based on the gold standard test (PCR).
Ratio of asymptomatic immunized (IgG) population | 2 months
  Statistical quantification of the rate of immunized (IgG) individuals attending to IVF clinics in the USA based on the ELISA test.

SECONDARY OUTCOMES:
To validate saliva specimens as a biological sample for COVID-19 testing | 2 months
  To validate the use of saliva specimen as a possible substitute to nasopharyngeal swabs, offering a simpler, easily self-sampling and large-scale test.

OTHER OUTCOMES:
Description of demographic characteristics | 2 months
  Age, gender and location distribution of affected contagious individuals in two areas of the USA with different pandemic status.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Cuzzi, PhD, Principal Investigator — Igenomix; Carlos Simon, MD, PhD, Principal Investigator — Igenomix
Locations (2):
- United States (2):
  - Boston IVF Fertility Clinic, Boston, Massachusetts
  - Utah Fertility Clinic, Pleasant Grove, Utah

IPD SHARING:
Plan to Share IPD: No